CLINICAL TRIAL: NCT07023562
Title: Comparing the Sample Quality of 22G Trident Needle Combined With Different Aspiration Techniques in EUS-Guided Fine-Needle Biopsy of Pancreatic Solid Lesions: A Randomized Controlled Multicenter Clinical Study
Brief Title: The 22G Trident Needle Combined With Different Aspiration Techniques for Endoscopic Ultrasound-guided Fine-needle Biopsy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Changhai Hospital (Other)
Responsible Party: Principal Investigator, Zhaoshen Li, Department of Gastroenterology, Changhai Hospital, Changhai Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: KTSB20250423035
Record Dates: First submitted 2025-06-08; First posted 2025-06-17 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Pancreatic Diseases
Keywords: EUS-FNB; solid pancreatic lesion; sample processing
MeSH Terms: conditions — Pancreatic Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ABC group (Experimental)
  Interventions: Procedure: ABC suction sequence
- ACB group (Experimental)
  Interventions: Procedure: ACB suction sequence
- BAC group (Experimental)
  Interventions: Procedure: BAC suction sequence
- BCA group (Experimental)
  Interventions: Procedure: BCA suction sequence
- CAB group (Experimental)
  Interventions: Procedure: CAB suction sequence
- CBA group (Experimental)
  Interventions: Procedure: CBA suction sequence

INTERVENTIONS:
Procedure: ABC suction sequence — Suction sampling should be conducted in the sequence of dry-suction, slow-pull and wet-suction.
  Arms: ABC group
Procedure: ACB suction sequence — Suction sampling should be conducted in the sequence of dry-suction, wet-suction and slow-pull.
  Arms: ACB group
Procedure: BAC suction sequence — Suction sampling should be conducted in the sequence of slow-pull, dry-suction and wet-suction.
  Arms: BAC group
Procedure: BCA suction sequence — Suction sampling should be conducted in the sequence of slow-pull, wet-suction and dry-suction.
  Arms: BCA group
Procedure: CAB suction sequence — Suction sampling should be conducted in the sequence of wet-suction, dry-suction and slow-pull.
  Arms: CAB group
Procedure: CBA suction sequence — Suction sampling should be conducted in the sequence of wet-suction, slow-pull and dry-suction.
  Arms: CBA group

SUMMARY:
The goal of this clinical study is to compare the tissue adequacy, cellularity, blood contamination, accuracy, sensitivity, specificity of the 22G Trident needle combined with three different aspiration techniques (dry-suction, wet-suction, and slow-pull) in Endoscopic ultrasound-guided fine-needle biopsy for solid pancreatic lesions.

DETAILED DESCRIPTION:
Patients who met the inclusion criteria of this trial and did not meet the exclusion criteria were randomly divided into six groups according to the crossover grouping design. Samples were collected using a 22G Trident needle in different suction sequences. The advantages and disadvantages of different suction techniques in terms of sample quality and diagnostic efficacy were compared to further clarify the optimal suction sampling scheme for Endoscopic ultrasound-guided fine-needle biopsy (EUS-FNB) using a 22G Trident needle.

ELIGIBILITY:
Inclusion Criteria:

* (Before the trial, subjects must meet all of the requirements listed below in order to be enrolled)

  1. 18-80 years old (inclusive), male and female;
  2. patients with pancreatic solid mass > 1cm detected by CT/MRI/PET-CT or EUS and requiring EUS-FNB diagnosis.
  3. written informed consent was obtained.

Exclusion Criteria:

* (Before the trial, participants could not be enrolled if they met any of the following requirements)

  1. contraindications to endoscopy, such as severe cardiovascular and cerebrovascular diseases;
  2. bleeding coagulation dysfunction (prothrombin international normalized ratio ≥1.5, platelet count ≤ 50 000) or use of antiplatelet drugs;
  3. confirmed pregnancy or possible pregnancy;
  4. pathological diagnosis has been obtained by other methods;
  5. refuse to participate in the study, are participating in another observational clinical trial, or have participated in another clinical trial within 60 days.
  6. other situations where EUS-FNB could not be performed.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-06-25 (Estimated); Primary Completion 2027-05-26 (Estimated); Study Completion 2027-05-26 (Estimated)

PRIMARY OUTCOMES:
Tissue adequacy | 2 months
  Grade A, existing core tissue (defined as structurally intact tissue with a long axis length of at least 550 μm) that clearly characterizes the lesion and is sufficient for diagnosis; Grade B, the presence of core fragments that do not meet the histological criteria for structural integrity, but can still be diagnosed based on cell morphology; Grade C, no diseased tissue is found and no diagnosis can be made based on the sample.

SECONDARY OUTCOMES:
Cellularity | 2 months
  Grade A: Satisfactory, with more than 4 clusters, each containing at least 10 cells for cytological analysis; Grade B: Adequate, with 2-4 clusters, each containing at least 10 cells for cytological analysis; Grade C: Insufficient, with<2 clusters suitable for cytological analysis or non-representative samples, or<50 cells with clear nuclear structures.
Blood contamination | 2 months
  The histological blood contamination score is assessed by grading the percentage of red blood cells in the entire 40x magnified field of view. Grade A: Red blood cells are present in<25%of the slides; Grade B: Red blood cells occupy 25%-50%of the slide; Grade C: Red blood cells are present in>50%of the slides; Grade D: No tissue.
Diagnostic accuracy | 6 months
  Diagnostic accuracy was calculated as the proportion of true positive and true negative in all evaluated cases.
Diagnostic sensitivity | 6 months
  Diagnostic sensitivity was calculated as the proportion of true positives in patient cases.
Diagnostic specificity | 6 months
  Diagnostic specificity was calculated as proportion of true negative in healthy cases.

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Shen Li, M.D, Principal Investigator — Department of Gastroenterology, Changhai Hospital, Naval Medical University (Second Military Medical University), shanghai, China
Locations (1):
- Changhai Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No